CLINICAL TRIAL: NCT07277712
Title: A Randomized, Open-label, Crossover Study to Evaluate the Pharmacokinetics Following Administration of IN-M00002 Tablet and Co-administration of Tegoprazan and Naproxen, and to Evaluate Food-effect of IN-M00002 Tablet in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Food-effect of IN-M00002 Tablet in Healthy Adult Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_TNA_101
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer
Keywords: pharmacokinetic; food-effect
MeSH Terms: interventions — tegoprazan; Naproxen

STUDY DESIGN:
Intervention Model Description: [Part A] 2-sequence-arm, 2-period crossover study [Part B] 2-sequence-arm, 2-period crossover study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Sequence 1 (Treatment A - Treatment B) (Experimental): Period 1: Single dose of tegoprazan 25 mg QD in combination with naproxen 500 mg BID Period 2: Single dose of IN-M00002 tablet BID
  Interventions: Drug: Tegoprazan; Drug: Naproxen; Drug: IN-M00002
- Part A: Sequence 2 (Treatment B - Treatment A) (Experimental): Period 1: Single dose of IN-M00002 tablet BID Period 2: Single dose of tegoprazan 25 mg QD in combination with naproxen 500 mg BID
  Interventions: Drug: Tegoprazan; Drug: Naproxen; Drug: IN-M00002
- Part B: Sequence 1 (Treatment C - Treatment D) (Experimental): Period 1: Single dose of IN-M00002 tablet QD under fasted conditions Period 2: Single dose of IN-M00002 tablet QD under fed conditions
  Interventions: Drug: IN-M00002
- Part B: Sequence 2 (Treatment D - Treatment C) (Experimental): Period 1: Single dose of IN-M00002 tablet QD under fed conditions Period 2: Single dose of IN-M00002 tablet QD under fasted conditions
  Interventions: Drug: IN-M00002

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 25 mg QD
  Other Names: K-CAB
  Arms: Part A: Sequence 1 (Treatment A - Treatment B); Part A: Sequence 2 (Treatment B - Treatment A)
Drug: Naproxen — Naproxen 500 mg BID
  Other Names: Naxen-F
  Arms: Part A: Sequence 1 (Treatment A - Treatment B); Part A: Sequence 2 (Treatment B - Treatment A)
Drug: IN-M00002 — IN-M00002 tablet QD
  Arms: Part B: Sequence 1 (Treatment C - Treatment D); Part B: Sequence 2 (Treatment D - Treatment C)
Drug: IN-M00002 — IN-M00002 tablet BID
  Arms: Part A: Sequence 1 (Treatment A - Treatment B); Part A: Sequence 2 (Treatment B - Treatment A)

SUMMARY:
This study aims to evaluate the pharmacokinetic (PK) following administration of IN-M00002 tablet and co-administration of tegoprazan and naproxen, and to evaluate food-effect of IN-M00002 tablet in healthy adult volunteers

DETAILED DESCRIPTION:
A randomized, open-label, crossover study

[Part A] To evaluate and compare the pharmacokinetic and safety of co-administration of tegoprazan and naproxen versus administration of IN-M00002 tablet in healthy adult volunteers

[Part B] To evaluate the effects of food on the pharmacokinetic and safety of IN-M00002 tablet in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged ≥ 19 and ≤ 55 year-old at screening
* Body mass index (BMI) ≥ 19.0 kg/m2 and ≤ 27.0 kg/m2 with a body weight ≥ 45 kg at screening
* Those determined to be eligible for this study based on the findings of screening such as clinical laboratory tests (hematological test, blood chemistry test, blood coagulation test, urinalysis, test for viruses/bacteria, etc.), vital signs, and electrocardiogram (ECG) which are performed by the investigator according to the properties of medicines
* Those who have fully understood this clinical trial via detailed explanation, were willing to voluntarily participate in this study, and agreed to give written informed consent prior to the screening
* Those with a capability/willingness to participate throughout the study

Exclusion Criteria:

* Medical history or evidence of clinically significant blood, renal, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological, musculoskeletal, oncological, or immune disease (except for history of simple dental treatment such as tartar, impacted teeth, and third molar teeth)
* Previous history of gastrointestinal disease (esophageal disease such as esophageal achalasia or esophageal stricture, inflammatory bowel disease (Crohn's disease, ulcerative colitis)) or surgery (except for simple appendectomy, hernia surgery, tooth extraction, etc.) which may affect drug absorption
* Sitting systolic blood pressure < 90 mmHg or ≥ 140 mmHg or diastolic blood pressure < 60 mmHg or ≥ 90 mmHg at screening
* Following findings of clinical laboratory tests:

  * ALT or AST value > twice the upper limit of normal (ULN)
* History of periodic alcohol consumption exceeding 210 g/week within 6 months prior to screening (beer (5%) 1 glass (250 mL) = 10 g, soju (20%) 1 glass (50 mL) = 8 g, wine (12%) 1 glass (125 mL) = 12 g)
* Has taken any other investigational product within 6 months prior to the first dose of investigational product
* History of serious alcohol or drug misuse and abuse within 1 year prior to screening
* Administration of drugs known to markedly induce or inhibit drug metabolizing enzymes within 30 days prior to the first dose of the investigational product
* Daily use of ≥ 20 cigarettes within 6 months prior to screening
* Administration of a prescription or non-prescription drug within 10 days prior to the first dose of the investigational product
* Whole blood donation within 2 months prior to the first dose of the investigational product or apheresis donation within 1 month prior to the first dose of the investigational product
* Subjects who received a blood transfusion within 1 month prior to the first dose of the investigational product
* Those who may be put at an increased risk due to the administration of the investigational product and study participation or have a severe acute/chronic medical or mental condition which may interfere with the interpretation of study results
* Subjects with a history of hypersensitivity (e.g., asthma, rhinitis, nasal polyps, urticaria, or allergic reactions) to the components of tegoprazan or naproxen, benzimidazole derivatives, aspirin, or other non-steroidal anti-inflammatory drugs (including COX-2 inhibitors)
* Subjects currently receiving medications containing atazanavir, nelfinavir, or rilpivirine
* Women with a positive pregnancy test, pregnant, or breastfeeding
* Subjects are unable to use a highly effective method of contraception (e.g., correctly placed intrauterine device(IUD), sterilization surgery (vasectomy, tubal ligation, etc.))
* Subjects unable to consume a high-fat diet provided during Part B of the clinical trial
* Subjects who are considered ineligible to participate in this study at the discretion of the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
AUCt of tegoprazan | Up to 48 hours
  Area under the plasma concentration-time curve from the time of dosing to the time of the last measurable concentration
AUCt of naproxen | Up to 72 hours
  Area under the plasma concentration-time curve from the time of dosing to the time of the last measurable concentration
Cmax of tegoprazan | Up to 48 hours
  Maximum plasma concentration of tegoprazan
Cmax of naproxen | Up to 72 hours
  Maximum plasma concentration of naproxen

CONTACTS AND LOCATIONS:
Overall Officials: Seol Ju Moon, MD, Ph.D, Principal Investigator — Clinical Pharmacology Center, Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea